CLINICAL TRIAL: NCT00508573
Title: Registry for Women Who Are At Risk Or May Have Lynch Syndrome
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0973
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hereditary Nonpolyposis Colorectal Cancer; Lynch Syndrome
Keywords: Hereditary Nonpolyposis Colorectal Cancer; Lynch Syndrome; HNPCC; Syndrome Registry; Questionnaire; Endometrial cancer; Ovarian cancer
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms; Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leftover tissue samples will be collected from surgery performed. These samples will be stored and used to perform molecular studies to characterize Lynch syndrome tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lynch Syndrome Registry: Patient that has or is at risk for Lynch Syndrome.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Follow-up questionnaire done once a year for five years.
  Other Names: Survey

SUMMARY:
The goal of this study is to create a registry of information about women who have or are at risk for Lynch syndrome, in order to study gynecologic cancer risks.

This is an investigational study. Up to 1000 patients will take part in this study. All patients will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Lynch Syndrome:

In women with hereditary non-polyposis colorectal cancer syndrome (HNPCC), also called Lynch syndrome, the lifetime risk for endometrial cancer increases to 40-60%, and the risk for ovarian cancer increases to 12%.

Study Procedures:

If you agree to take part in this study, basic medical and family information will be collected. You will be asked to fill out a baseline (starting) questionnaire, which will ask personal information such as age, ethnic background, medical and family history, and health habits. All information will be kept confidential. Some information may be gathered from your medical record. It should take about 30 minutes to complete this questionnaire.

Once a year for 20 years, you will be asked to complete a follow-up questionnaire. The follow-up questionnaire provides researchers with an opportunity to study possible health issues and/or changes that may have occurred since your last visit. This questionnaire should only take about 15 -20 minutes to complete.

If you have a history of endometrial or ovarian cancer, or develop endometrial or ovarian cancer while on study, researchers will collect copies of the diagnostic and surgery reports from your medical record and will ask you to fill out an additional questionnaire about symptoms of endometrial cancer. This should only take about 15 minutes to complete.

Researchers will also collect several leftover tissue samples from your surgery if you have had surgery. These samples will be stored and used to perform molecular studies to characterize Lynch syndrome tumors. The samples will be kept securely in a lab at MD Anderson.

Before your leftover tissue samples can be used for research, the people doing the research must get specific approval from the Institutional Review Board (IRB) of MD Anderson. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at MD Anderson, including research involving your leftover tissue samples must first be approved by the IRB.

Length of Study:

At the end of the study, you may be invited to participate in a follow-up study. During your participation in this registry study, researchers will inform you about related studies for which you might be eligible. You will have the option to take part or not to take part in them. Your active participation in this study will continue for up to 20 years total.

ELIGIBILITY:
Inclusion Criteria:

1. Women who meet one or more of the following criteria : A.Lynch syndrome mutation, including those at risk for cancer, those who have had cancer, and those who have had prophylactic surgery. B. Family history meets Amsterdam II criteria, defined as the following: At least 3 relatives with an HNPCC-associated cancer (colorectal.endometrial cancer, small bowel, ureter, or renal pelvis).One is a first-degree relative of the other two. At least 2 successive generations affected. One cancer diagnosed before age 50.C. Tumor studies (MSI, IHC) are suggestive for Lynch Syndrome.
2. D. Female family members who are at 25% or 50% risk for a lynch syndrome mutation may also be enrolled in the registry. 25% risk is defined as women with second degree family member grandmother, aunt, uncle, niece, and grandchild. 50% risk is defined as women with first degree family member being parent, child, sibling.
3. Subjects must be 18 or older and able to give informed consent.

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, 18 years or older, that have or are at risk for Lynch Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Number of Women Participating in Registry | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org